CLINICAL TRIAL: NCT05316129
Title: A Phase I Clinical Trial of an Infusion of Autologous T Cells Genetically Engineered With a Chimeric Receptor to Target the Follicle-Stimulating Hormone Receptor in Patients With Recurrent Ovarian Cancer
Brief Title: Infusion of Autologous T Cells Engineered to Target FSH Receptor in Recurrent Ovarian Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Anixa Biosciences, Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MCC-21113
Record Dates: First submitted 2022-03-30; First posted 2022-04-07 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (10):
- Intraperitoneal treatment- Dose Level 1 (Experimental): Participants will receive one infusion of Follicle-Stimulating Hormone Receptor T (FSHCER T) cells at a dose of 1 x 10^5. Intraperitoneal: Infusion will be administered through a thin membrane of the abdominal cavity.
  Interventions: Drug: Follicle Stimulating Hormone Receptor T Cells
- Intravenous treatment - Dose Level 1 (Experimental): Participants will receive one infusion of Follicle-Stimulating Hormone Receptor T (FSHCER T) cells at a dose of 1 x 10^5 by Intravenous (IV).
  Interventions: Drug: Follicle Stimulating Hormone Receptor T Cells
- Intraperitoneal treatment- Dose Level 2 (Experimental): Participants will receive one infusion of Follicle-Stimulating Hormone Receptor T (FSHCER T) cells at a dose of 3 x 10^5. Intraperitoneal: Infusion will be administered through a thin membrane of the abdominal cavity.
  Interventions: Drug: Follicle Stimulating Hormone Receptor T Cells
- Intravenous treatment - Dose Level 2 (Experimental): Participants will receive one infusion of Follicle-Stimulating Hormone Receptor T (FSHCER T) cells at a dose of 3 x 10^5 by Intravenous (IV).
  Interventions: Drug: Follicle Stimulating Hormone Receptor T Cells
- Intraperitoneal treatment- Dose Level 3 (Experimental): Participants will receive one infusion of Follicle-Stimulating Hormone Receptor T (FSHCER T) cells at a dose of 1 x 10^6. Intraperitoneal: Infusion will be administered through a thin membrane of the abdominal cavity.
  Interventions: Drug: Follicle Stimulating Hormone Receptor T Cells
- Intravenous treatment - Dose Level 3 (Experimental): Participants will receive one infusion of Follicle-Stimulating Hormone Receptor T (FSHCER T) cells at a dose of 1 x 10^6 by Intravenous (IV).
  Interventions: Drug: Follicle Stimulating Hormone Receptor T Cells
- Intraperitoneal treatment- Dose Level 4 (Experimental): Participants will receive one infusion of Follicle-Stimulating Hormone Receptor T (FSHCER T) cells at a dose of 3 x 10^6. Intraperitoneal: Infusion will be administered through a thin membrane of the abdominal cavity.
  Interventions: Drug: Follicle Stimulating Hormone Receptor T Cells
- Intravenous treatment - Dose Level 4 (Experimental): Participants will receive one infusion of Follicle-Stimulating Hormone Receptor T (FSHCER T) cells at a dose of 3 x 10^6 by Intravenous (IV).
  Interventions: Drug: Follicle Stimulating Hormone Receptor T Cells
- Intraperitoneal treatment- Dose Level 5 (Experimental): Participants will receive one infusion of Follicle-Stimulating Hormone Receptor T (FSHCER T) cells at a dose of 1 x 10^7. Intraperitoneal: Infusion will be administered through a thin membrane of the abdominal cavity.
  Interventions: Drug: Follicle Stimulating Hormone Receptor T Cells
- Intravenous treatment - Dose Level 5 (Experimental): Participants will receive one infusion of Follicle-Stimulating Hormone Receptor T (FSHCER T) cells at a dose of 1 x 10^7 by Intravenous (IV).
  Interventions: Drug: Follicle Stimulating Hormone Receptor T Cells

INTERVENTIONS:
Drug: Follicle Stimulating Hormone Receptor T Cells — Participants will receive an infusion of autologous t cells genetically modified ex vivo to express the FSHR-specific 4-1BB/CD3ζ CER.

SUMMARY:
The purpose of this first in human study is to evaluate the safety of treatment with autologous T cells genetically modified to express a CER (chimeric endocrine receptor) targeting the FSHR (follicle-stimulating hormone receptor) (FSHCER T cells), with or without conditioning chemotherapy, in participants with recurrent or persistent ovarian, fallopian tube, or primary peritoneal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older and able to provide informed consent.
* Pathologically confirmed diagnosis of invasive (Grades 1-3) epithelial ovarian cancer, primary peritoneal cancer, or fallopian tube carcinoma (EOC), which are serous, endometrioid, clear cell, mucinous, mixed epithelial, or undifferentiated. Borderline serous ovarian tumors (BOT, also known as serous low-malignant potential tumors) are included, as are mixed invasive/borderline cancers. Patients may also have sex cord-stromal tumors (SCSTs) to include adult-type granulosa cell tumors (GCTs) and Sertoli Leydig cell tumors (SLCTs), or SCSTs with mixed elements that include at least one of these types.
* Have measurable disease or detectable (non-measurable) disease.
* Consent to have tumor obtained for correlative study testing.
* Patients must have had 1 prior platinum-based chemotherapeutic regimen for the management of ovarian, primary peritoneal, or fallopian tube carcinoma and at least 2 prior chemotherapy regimens.
* Patients should be considered platinum- refractory (progression while on a prior platinum chemotherapy) or resistant (persistence or recurrence within 6 months after a prior platinum chemotherapy) and be deemed unlikely to have significant benefit from any standard therapies by the treating investigator.
* Patients with a known germline or somatic BRCA pathogenic mutation should receive a PARP inhibitor if treatment would be consistent with the current FDA approval for use of PARPi at time of screening, unless they have a documented history of intolerance or inability to swallow oral medications.
* For Granulosa Cell Tumors (GCTs), at least one hormonal regimen (i.e., letrozole) should be included in prior therapies.
* For Borderline Ovarian Tumors, documentation of the consideration of a MEK inhibitor (e.g., trametinib) should be included.
* For high-grade serous (Grades 2,3), eligibility and consideration of Folate Receptor-alpha antibody drug conjugate (e.g., mirvetuxumab) should be considered and documented for patients who meet all FDA label criteria.
* Patients are allowed to receive, but are not required to receive, up to 6 additional prior (for a total of 8 prior treatments) chemotherapy treatment regimens (including platinum-based chemotherapy). Prior maintenance therapy with an agent when there has not been progression will not be a separate treatment regimen. Prior hormonal therapy is allowed, and when used alone, even as a therapeutic agent, it does not count toward this prior regimen requirement. Hormonal therapy must be discontinued at least 1 week before T-cell infusion. Continuation of hormone replacement therapy is permitted.
* Patients are allowed to receive, but are not required to receive, biologic/targeted therapy alone or as part of their treatment regimens. When used as treatment after progression, these treatments will count as a separate therapy.
* Eastern Cooperative Oncology Group (ECOG) status of 2 or better (or Karnofsky Performance Status score of ≥60%).
* Life expectancy of at least 3 months.
* Adequate bone marrow, renal, and hepatic function (liver function and renal tests, grade 1 or lower):
* No anticancer therapy (chemotherapy, biologic therapy, or immunotherapy) in the 3 weeks before the T-cell infusion (and all hematologic effects have resolved).
* No prior immunotherapy with checkpoint blockade (e.g., PD1 inhibitor, PDL1 inhibitor, or CTL4- antagonist or similar agent) in the 3 months before the T-cell infusion (and all clinically significant related side effects must be resolved).
* Patient agrees to undergo placement of surgically placed peritoneal port and central line catheter. (may be temporary or subcutaneous).
* Although it is anticipated that patients who are eligible for this study will not have childbearing potential, any patient the treating doctor or investigator deems to have childbearing potential must agree to an acceptable means of contraception from the time of screening to at least 6 months after T-cell infusion.

Exclusion Criteria:

* Known active hepatitis B infection, known history of hepatitis C or HIV infection.
* Clinical or radiographic evidence of bowel obstruction or need for parenteral hydration and/or nutrition.
* Known or suspected extensive abdominal adhesions that would preclude port placement or infusion.
* Any of the following cardiac conditions:

Clinically significant heart disease (New York Heart Association class 3 or 4) or symptomatic congestive heart failure.

Myocardial infarction <6 months before enrollment. History of clinically significant ventricular arrhythmia or unexplained syncope that is not believed to be vasovagal in nature or due to dehydration.

History of severe non-ischemic cardiomyopathy with ejection fraction <20%. Findings on baseline ECG or ECHO that, in the opinion of the patient's treating physician or investigator, would require medical intervention before anticancer therapy

* Active autoimmune disease (excluding autoimmune thyroid disease on a stable thyroid regimen). Such conditions include but are not limited to systemic lupus erythematous, rheumatoid arthritis, ulcerative colitis, Crohn's disease, and temporal arteritis.
* Known or suspected leptomeningeal disease and patients with metastases to the brain stem, midbrain, pons, or medulla.
* Known or suspected untreated brain metastases. Patients with radiographically stable, asymptomatic previously irradiated lesions are eligible provided patient is >4 weeks beyond completion of cranial irradiation and >3 weeks off of corticosteroid therapy at the time of study intervention.
* Prior history of clinically significant seizure disorder (e.g., not including childhood febrile seizures).
* Any concurrent active malignancies, defined as malignancies requiring any therapy other than expectant observation, because adverse events (AEs) resulting from these malignancies or their treatment may confound our assessment of the safety of adoptive T-cell therapy for ovarian cancer.
* Prior radiotherapy to any portion of the abdominal cavity or pelvis.
* Current lactation or pregnancy
* Any of the following within 28 days of first date of study treatment:

Serious uncontrolled medical illness or disorder that in the opinion of the treating physician would make the patient ineligible for the study.

Active uncontrolled infection (with the exception of uncomplicated urinary tract infection).

Abdominal fistula, gastrointestinal perforation, or intraabdominal abscess. Abdominal surgery (for reasons other than IP port placement).

* Any other issue which, in the opinion of the treating physician or principal investigator, would make the patient ineligible for the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — female participants only
Enrollment: 10 (Estimated)
Dates: Start 2022-04-28 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2029-05 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose of FSHCER T Cells | Day 1
  Participants will receive escalating doses of FSHCER T Cells to determine the Maximum Tolerated Dose (MTD). MTD is defined as the the highest dose of t cells that does not cause unacceptable side effects.

SECONDARY OUTCOMES:
Duration of Response | Up to 15 years
  The duration of response is measured from the time measurement criteria are met for immune complete response or immune partial response (whichever is first recorded) until the first date that progressive disease (immune related progressive disease -irPD) is objectively documented (taking as reference for PD the smallest measurements recorded [nadir] since the treatment started).
Duration of Stable Disease | Up to 15 years
  Stable Disease is measured from the start of the treatment until the criteria for confirmed progressive disease are met.
Overall Survival | Up to 15 years
  Overall survival defined as the time from initial date of treatment to date of death.

CONTACTS AND LOCATIONS:
Overall Officials: Robert M Wenham, MD, MS, FACOG, FACS, Principal Investigator — Moffitt Cancer Center
Locations (1):
- Moffitt Cancer Center, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided